CLINICAL TRIAL: NCT03545841
Title: High-Intensity Interval Training Improves Aerobic Capacity and Abolishes the Decline in Blood Glucose Observed During Moderate-Intensity Continuous Training Sessions in People With Type 1 Diabetes
Brief Title: HIT in People With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Sam Shepherd, Dr Sam Shepherd, Principle Investigator, Liverpool John Moores University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: T1D_PARTB
Record Dates: First submitted 2018-05-09; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIT training (Experimental): 6 weeks of high-intensity interval training (HIT)
  Interventions: Other: HIT
- Moderate intensity training (Experimental): 6 weeks of moderate-intensity continuous training (MICT)
  Interventions: Other: MICT

INTERVENTIONS:
Other: HIT — Participants completed 6 weeks of HIT
  Arms: HIT training
Other: MICT — Participants completed 6 weeks of MICT
  Arms: Moderate intensity training

SUMMARY:
Few people with type 1 diabetes achieve exercise guidelines and many programmes designed to increase physical activity have failed. High-intensity interval training (HIT) has been shown to be a time-efficient alternative to traditional moderate-intensity continuous training (MICT) in various groups without type 1 diabetes. A single bout of HIT does not increase the risk of hypoglycaemia in people with type 1 diabetes. This study aimed to assess whether HIT a safe, effective and time-efficient training strategy to improve cardio-metabolic health and reduce the risk of hypoglycaemia in people with type 1 diabetes.

DETAILED DESCRIPTION:
This study aimed to investigate whether 1) six weeks of high-intensity interval training (HIT) induces similar improvements in cardio-metabolic health markers as moderate-intensity continuous training (MICT) in people with type 1 diabetes, and 2) whether HIT abolishes acute reductions in plasma glucose observed following MICT sessions. Fourteen sedentary individuals with type 1 diabetes (n=7 per group) completed six weeks of HIT or MICT 3 times per week. Pre- and post-training measurements were made of 24h interstitial glucose profiles (using continuous glucose monitors (CGMS)) and cardio-metabolic health markers (V ̇O2peak, blood lipid profile and aortic pulse wave velocity; aPWV). Capillary blood glucose concentrations were assessed before and after exercise sessions throughout the training programme to investigate changes in blood glucose during exercise in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes >6 months
* basal bolus regimen
* no significant history of hyper- or hypoglycaemia (determined from medical history)

Exclusion Criteria:

duration of type 1 diabetes <6 months,

* insulin pump therapy
* significant history of hyper- or hypoglycaemia (determined from medical history)
* obesity (BMI >30 kg∙m-2)
* pregnancy or planning pregnancy
* uncontrolled hypertension (>180/100 mmHg)
* angina, autonomic neuropathy
* taking any medication that affects heart rate
* major surgery planned within 6 weeks of the study
* severe nonproliferative
* unstable proliferative retinopathy

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Maximal aerobic capacity | change in baseline maximal aerobic capacity at 6 weeks
  Maximal aerobic capacity test pre and post 6-week training intervention

SECONDARY OUTCOMES:
Vascular stiffness | change in baseline vascular stiffness at 6 weeks
  Aortic pulse wave velocity to measure vascular stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to make data available to others